CLINICAL TRIAL: NCT06988501
Title: The Effect of Goal Setting With Mobile-based Self-management Tool on Improving Diet Quality of People With High Blood Pressure: a Randomized Controlled Trial
Brief Title: Goal Setting and Mobile-based Self-management Tool to Improve Diet Quality of People With High Blood Pressure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-2167
Record Dates: First submitted 2025-05-16; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2024-10

CONDITIONS: Blood Pressure, High
Keywords: goal setting
MeSH Terms: conditions — Hypertension | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group will receive nutrition education on blood pressure management. The dietitian will work with the participants to set individual SMART goals. The participants will have access to diet tracking function, weekly reports and monthly virtual meeting with dietitian.
  Interventions: Behavioral: Goal setting with mobile-based self-management tool
- Control group (Active Comparator): The control group will receive nutrition education on blood pressure management.
  Interventions: Other: Nutrition education

INTERVENTIONS:
Behavioral: Goal setting with mobile-based self-management tool — In addition to the nutrition education provided to both groups, the participants of the intervention group will work with the dietitian to make behavior-change goals based on SMART goal setting strategy. They will also have access to diet tracking function and weekly report on smart phone application. The dietitian will also meet with the participants virtually to track their progress and provide suggestions.
  Arms: Intervention group
Other: Nutrition education — The control group will receive nutrition education about blood pressure management by the dietitian
  Arms: Control group

SUMMARY:
SMART goal setting is a patient-led method that can help improve execution and facilitate behavioral changes. Functions such as diet tracking, interaction, and feedback in smartphone application may help enhance patient compliance. This study aims to explore the nutrition intervention measures of SMART goal setting combined with smartphone applications for daily self-management on the effect of improving diet quality of people with high blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-70;
* Hypertension diagnosis, or high blood pressure (SBP between 120-139 mmHg and/or DBP between 80-89 mmHg);
* Eating an unhealthy diet (estimated DASH score < 6) ;
* Owning a smartphone and able to operate it proficiently;
* Sign the informed consent.

Exclusion Criteria:

* Severe cardiovascular and respiratory diseases, such as acute myocardial infarction, tachyarrhythmia, pulmonary edema, and severe aortic stenosis;
* Acute phase of cardiovascular and cerebrovascular diseases;
* Uncontrolled blood pressure;
* Diagnosed mental diseases or epilepsy;
* Cardiac pacemaker implantation;
* Allergic constitutions;
* Pregnant women or planning to become pregnant;
* Individuals who have participated in other clinical studies within the past 3 months;
* Refuse to sign the informed consent.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-07-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Diet quality | From enrollment to the end of treatment at 12 weeks
  Diet quality is measured by the DASH Score that includes eight dietary components to reflect the adherence to the DASH dietary pattern.

SECONDARY OUTCOMES:
Blood pressure | From enrollment to the end of treatment at 12 weeks
  Blood pressure will be measured at baseline visit and the follow-up visit after the 12-week intervention. Blood pressure will be measured using calibrated electronic blood pressure monitor.
Body Weight | From enrollment to the end of treatment at 12 weeks
  Body weight will be measured by the bioelectrical impedance analysis.

OTHER OUTCOMES:
Sleep Quality | From enrollment to the end of treatment at 12 weeks
  Sleep quality will be measured by the Pittsburgh Sleep Quality Index
Depression | From enrollment to the end of treatment at 12 weeks
  Depressive status will be measured by the Patient Health Questionnaire-9
Anxiety | From enrollment to the end of treatment at 12 weeks
  Anxiety status will be measured by the Generalized Anxiety Disorder-7.

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital, National Center for Cardiovascular Diseases, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kassavou A, Wang M, Mirzaei V, Shpendi S, Hasan R. The Association Between Smartphone App-Based Self-monitoring of Hypertension-Related Behaviors and Reductions in High Blood Pressure: Systematic Review and Meta-analysis. JMIR Mhealth Uhealth. 2022 Jul 12;10(7):e34767. doi: 10.2196/34767. PMID 35819830
- [Background] Villinger K, Wahl DR, Boeing H, Schupp HT, Renner B. The effectiveness of app-based mobile interventions on nutrition behaviours and nutrition-related health outcomes: A systematic review and meta-analysis. Obes Rev. 2019 Oct;20(10):1465-1484. doi: 10.1111/obr.12903. Epub 2019 Jul 28. PMID 31353783
- [Background] Limketkai BN, Mauldin K, Manitius N, Jalilian L, Salonen BR. The Age of Artificial Intelligence: Use of Digital Technology in Clinical Nutrition. Curr Surg Rep. 2021;9(7):20. doi: 10.1007/s40137-021-00297-3. Epub 2021 Jun 8. PMID 34123579
- [Background] White ND, Bautista V, Lenz T, Cosimano A. Using the SMART-EST Goals in Lifestyle Medicine Prescription. Am J Lifestyle Med. 2020 Feb 17;14(3):271-273. doi: 10.1177/1559827620905775. eCollection 2020 May-Jun. PMID 32477026
- [Background] Wing RR, Jeffery RW. Benefits of recruiting participants with friends and increasing social support for weight loss and maintenance. J Consult Clin Psychol. 1999 Feb;67(1):132-8. doi: 10.1037//0022-006x.67.1.132. PMID 10028217
- [Background] Boutelle KN, Kirschenbaum DS, Baker RC, Mitchell ME. How can obese weight controllers minimize weight gain during the high risk holiday season? By self-monitoring very consistently. Health Psychol. 1999 Jul;18(4):364-8. doi: 10.1037//0278-6133.18.4.364. PMID 10431937
- [Background] Mellen PB, Gao SK, Vitolins MZ, Goff DC Jr. Deteriorating dietary habits among adults with hypertension: DASH dietary accordance, NHANES 1988-1994 and 1999-2004. Arch Intern Med. 2008 Feb 11;168(3):308-14. doi: 10.1001/archinternmed.2007.119. PMID 18268173
- [Background] Yu D, Zhang X, Xiang YB, Yang G, Li H, Gao YT, Zheng W, Shu XO. Adherence to dietary guidelines and mortality: a report from prospective cohort studies of 134,000 Chinese adults in urban Shanghai. Am J Clin Nutr. 2014 Aug;100(2):693-700. doi: 10.3945/ajcn.113.079194. Epub 2014 Jun 18. PMID 24944055
- [Background] Savica V, Bellinghieri G, Kopple JD. The effect of nutrition on blood pressure. Annu Rev Nutr. 2010 Aug 21;30:365-401. doi: 10.1146/annurev-nutr-010510-103954. PMID 20645853
- [Background] Wang A, Tian X, Zuo Y, Chen S, Zhang Y, Zhang X, Deng X, Xu Q, Wang P, Wu S, Zhou Y. Control of Blood Pressure and Risk of Cardiovascular Disease and Mortality in Elderly Chinese: A Real-World Prospective Cohort Study. Hypertension. 2022 Aug;79(8):1866-1875. doi: 10.1161/HYPERTENSIONAHA.122.19587. Epub 2022 Jun 15. PMID 35706092
- [Background] Lewington S, Clarke R, Qizilbash N, Peto R, Collins R; Prospective Studies Collaboration. Age-specific relevance of usual blood pressure to vascular mortality: a meta-analysis of individual data for one million adults in 61 prospective studies. Lancet. 2002 Dec 14;360(9349):1903-13. doi: 10.1016/s0140-6736(02)11911-8. PMID 12493255
- [Background] Fuchs FD, Whelton PK. High Blood Pressure and Cardiovascular Disease. Hypertension. 2020 Feb;75(2):285-292. doi: 10.1161/HYPERTENSIONAHA.119.14240. Epub 2019 Dec 23. PMID 31865786